CLINICAL TRIAL: NCT04895293
Title: Evaluation of RBM-007 in Subjects With Treatment naïve Exudative Age-related Macular Degeneration (AMD)
Brief Title: RBM-007 in Treatment naïve Exudative Age-related Macular Degeneration
Acronym: TEMPURA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RKM-011
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: All subjects receive the study treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RBM-007 Injectable Solution - 2.0 mg (Experimental): Single intravitreal injection in study eye
  Interventions: Drug: RBM-007 Injectable Solution

INTERVENTIONS:
Drug: RBM-007 Injectable Solution — Sterile solution

SUMMARY:
This study is a single-center, open label, 4-month study, designed to evaluate the safety and treatment efficacy of RBM-007 in patients with intraretinal or subretinal edema due to previously untreated neovascular AMD. Up to 5 subjects will be randomized to receive study medication. Study treatment will be administered by intravitreal injections.

ELIGIBILITY:
Inclusion Criteria:

• General Inclusion Criteria:

1. Male or female patients, 50 years of age or older at baseline
2. Patient has completed/signed an informed consent prior to any study-related procedures and is able to follow study instructions and likely to complete all required visits.

   • Ocular Inclusion Criteria:
3. Best Corrected Visual Acuity (BCVA) 5 - 73 ETDRS letters (20/800-20/40 Snellen equivalent), inclusive, in study eye
4. Presence of choroidal neovascularization secondary to AMD
5. Clear ocular media and adequate pupil dilation to permit good quality photographic imaging.

Exclusion Criteria:

• General Exclusion Criteria:

1. Females who are pregnant, nursing, planning a pregnancy or who are of childbearing potential not using a reliable method of contraception.
2. History or current evidence of hypersensitivity to any components of the study medication or fluorescein, as assessed by the investigator.
3. Participation in any investigational drug or device study within 30 days prior to baseline
4. History or current evidence of a medical condition that may, in the opinion of the investigator, preclude the safe administration of study medication or affect the results of the study.

   • Ocular Exclusion Criteria:
5. Active ocular or periocular infections, malignancy
6. Aphakia
7. History of pars plana vitrectomy in the study eye
8. History of major ophthalmic surgery in the past 3 months in the study eye, or minor surgery in the past 30 days
9. History of significant ocular disease other than exudative AMD that may confound results
10. Uncontrolled glaucoma (defined as intraocular pressure >21mm Hg despite treatment with ocular hypotensive medications at baseline).

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K. Maturi, M.D., Study Chair — Midwest Eye Institute
Locations (1):
- Midwest Eye Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBM-007 Injectable Solution - 2.0 mg
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RBM-007 Injectable Solution - 2.0 mg
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Visual Acuity [Mean (Full Range); unit: Letters seen on eye chart] | 66.6 [57 to 73]
Central subfield thickness [Mean (Full Range); unit: Microns] | 422.8 [350 to 579]

OUTCOME MEASURES:

1. Primary Outcome: Macular Edema
Description: Central subfield thickness on optical coherence tomography
Time Frame: 3 months
Measure: Mean (Full Range); unit: Microns
Arm/Group | RBM-007 Injectable Solution - 2.0 mg
Number analyzed (Participants) | 5
Microns | 416 [257 to 648]

2. Secondary Outcome: Visual Acuity
Description: Change from Baseline in Best Corrected Visual Acuity
Time Frame: 3 Months
Measure: Mean (Full Range); unit: Letters seen on eye chart
Arm/Group | RBM-007 Injectable Solution - 2.0 mg
Number analyzed (Participants) | 5
Letters seen on eye chart | 60 [28 to 77]

ADVERSE EVENTS:
Time Frame: 3 months
Description: All adverse events and serious adverse events were continually assessed throughout the study. The investigator assessed safety throughout the study to determine appropriateness of continuing dosing and enrollment.
Arm/Group | RBM-007 Injectable Solution - 2.0 mg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBM-007 Injectable Solution - 2.0 mg (N=5)
Positive COVID test (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subretinal hemorrhage (Eye disorders) | 1 (1)
Myocardial infarction (mild) (Cardiac disorders) | 1 (1)
Diarrhea (severe) (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT04895293/Prot_SAP_000.pdf